CLINICAL TRIAL: NCT07016711
Title: Adherence to the Mediterranean Diet Among Women Attending Mammographic Screening in the "Prevention Caravan" by Komen Italy: a Cross-sectional Study
Brief Title: Adherence to the Mediterranean Diet Among Women Attending Mammographic Screening
Acronym: PREVCAR
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Boccia Stefania, Professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 7535
Record Dates: First submitted 2025-05-20; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer Prevention

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Lifestyle and Nutrition Promotion — Adherence to the Mediterranean diet

SUMMARY:
The PREVCAR study is a cross-sectional investigation aimed at evaluating dietary habits among women undergoing breast cancer screening. Specifically, the study focuses on adherence to the Mediterranean diet, a dietary pattern recognized for its potential protective role against chronic diseases, including breast cancer. The PREVCAR study will include approximately 35,000 women aged 18 and older who participate in the "Prevention Caravan" and complete both the breast cancer screening and the MEDAS (Mediterranean Diet Adherence Screener) questionnaire. This 14-item questionnaire measures dietary behavior, with scores reflecting levels of adherence to the Mediterranean diet.

The primary objective of the study is to determine the average MEDAS score among participants. Secondary objectives include analyzing how adherence varies across different known breast cancer risk factors-such as age, menopausal status, hormonal therapy use, and reproductive history-and assessing the prevalence of malignant breast lesions identified through the screening.

ELIGIBILITY:
Inclusion Criteria:

* Women who participate in the "Prevention Caravan" program;
* Women who undergo breast cancer screening, including mammography or breast ultrasound;
* Women who complete the MEDAS questionnaire.

Exclusion Criteria:

* Women who do not participate in the "Prevention Caravan" program;
* Women who participate in the "Prevention Caravan" program but undergo screenings or consultations for conditions other than breast cancer, such as gynecological cancers, thyroid ultrasounds, or dermatological evaluations;
* Women who do not complete the MEDAS questionnaire.

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: The study will focus on women aged 18 and older who will participate in mammographic screenings organized by the "Prevention Caravan" and who, due to age or other factors, are not eligible for breast cancer screening programs through the National Health Service (NHS). These screenings are primarily offered to women experiencing social or economic hardship, such as those living in suburban areas of Italian cities, women in detention, prison staff, and women residing in shelters. However, the program is also open to all women who exceed the age limits set by regional screening programs. Awareness of the "Prevention Caravan" program raises through advertising campaigns, making it accessible to a wider audience, and participants can easily register online. A total of 35,000 women will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 35000 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
Adherence to the MedDiet | At the moment of enrollment
  To assess adherence to the MedDiet, as measured by the Mediterranean Diet Adherence Screener (MEDAS) questionnaire, among women participating in mammographic screenings organized by the "Prevention Caravan" program. Adherence to the MedDiet was evaluated using the 14-item MEDAS questionnaire (S), a validated tool designed to assess specific dietary behaviors-including the consumption of olive oil, fruits, vegetables, legumes, fish, white meat, and wine-as well as the intake of foods considered inconsistent with the Mediterranean dietary pattern, such as red meat, butter, and sugar-sweetened beverages. Each item is scored as 0 or 1 based on the participant's response, resulting in a total score ranging from 0 to 14. Higher scores indicate greater adherence: scores above 10 are classified as excellent, scores between 8 and 10 as good, and scores below 8 as poor adherence to the MedDiet.

SECONDARY OUTCOMES:
MedDiet adherence levels across different categories of known breast cancer risk factors | At the moment of enrollment
  To assess the frequency of MedDiet adherence levels across different categories of known breast cancer risk factors
Malignant breast lesion | After 1 year, when women will be contact by phone to collect follow-up information on the outcomes of their breast screening
  The presence of malignant breast lesion in a subgroup of women participating in mammographic screenings